CLINICAL TRIAL: NCT04678323
Title: Improving Access to Anti-Obesity Pharmacotherapy for Pediatric Obesity: A Randomized Placebo-Controlled Trial of Phentermine
Brief Title: Pharmacotherapy for Pediatric Obesity: A Phentermine Clinical Trial
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPOM-P01
Record Dates: First submitted 2020-12-07; First posted 2020-12-21 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Obesity, Childhood
Keywords: Obesity
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Intervention Model Description: This study will randomize participants in a 1:1 manner to receive phentermine plus lifestyle therapy or placebo plus lifestyle therapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phentermine Plus Lifestyle Therapy (Active Comparator): Participants in this arm will receive 15 mg p.o.q.day of phentermine plus lifestyle therapy for 52 weeks.
  Interventions: Drug: Lifestyle Management
- Placebo Plus Lifestyle Therapy (Placebo Comparator): Participants in this arm will receive a matching placebo plus lifestyle therapy for 52 weeks.
  Interventions: Drug: Lifestyle Management

INTERVENTIONS:
Drug: Lifestyle Management — Participants in this group will receive lifestyle management.

SUMMARY:
This is a multi-site, randomized, placebo-controlled clinical trial to examine the weight loss efficacy and cardiovascular safety of phentermine 15 mg daily plus lifestyle therapy versus placebo plus lifestyle therapy among 200 adolescents ages ≥10 to <18 years with obesity.

DETAILED DESCRIPTION:
Obesity in children and adolescents (body mass index [BMI] ≥95th percentile) is a chronic, progressive, and debilitating disease with a prevalence of >20% in the U.S.1 Cardiovascular (CV) complications of obesity in this population are common,2 with nearly 40% of youth having ≥2 CV risk factors. Moreover, obesity in youth increases the risk of CV mortality in adulthood by nearly 5-fold. Treatment of obesity in adolescents includes lifestyle therapy (LST), and when this is ineffective, adjunct pharmacotherapy is recommended.5 However, there are few pharmacological options for pediatric obesity, and none are utilized to any significant degree by primary care pediatricians, even though obesity is the most common chronic disease of childhood.

Currently, orlistat is the only medication approved by the U.S. Food and Drug Administration (FDA) for the treatment of obesity in youth ages ≥12 years. However, adoption of orlistat in the clinical setting has been hampered by its significant side effects and poor accessibility due to high cost and poor insurance coverage. Two additional anti-obesity medications, liraglutide and combination phentermine-topiramate, are in the FDA approval pipeline for pediatric obesity, yet these are also unlikely to be widely prescribed by primary care pediatricians. Both of these medications are also expensive and are unlikely to be covered by many insurance plans. Furthermore, liraglutide is delivered by injection and topiramate has associated cognitive side effects. The paucity of safe, effective, and accessible pharmacological options has spurred pediatric obesity specialists to improvise by utilizing medications in an "off-label" manner, resorting to extrapolation of safety and efficacy data from adult clinical trials and opting for medications that are either covered by insurance or are inexpensive. One of the most commonly used medications prescribed in an "off-label" manner is phentermine.

Phentermine, a sympathomimetic, was FDA approved for obesity in 1959, before obesity was considered a chronic disease and when standards for clinical trials were lower than today. Accordingly, it was approved for short-term use, often interpreted as ≤12 weeks, in people ages >16 years. The popularity of phentermine among pediatric obesity specialists is likely driven by its demonstrated safety and efficacy in adults (4-5% mean placebo-subtracted weight loss over 26-28 weeks), oral route of administration, and affordability. Yet in spite of its popularity and routine use beyond 12 weeks, significant gaps exist in our knowledge regarding its safety and efficacy in children and adolescents, many of whom may have abnormal CV profiles at baseline. Indeed, pediatric data regarding phentermine use are sparse: only one retrospective clinical report (published by our group), demonstrated a 4% BMI reduction at 6 months with no significant increase in blood pressure.

To address these important gaps and generate evidence to directly inform clinical care, we propose this multi-site, randomized, placebo-controlled clinical trial to examine the weight loss efficacy and CV safety of phentermine 15 mg daily plus LST vs. placebo plus LST among 200 adolescents ages ≥10 to <18 years with obesity. To maximize the overall impact and clinical scalability, our explicit goal will be to generate the data necessary to support an FDA label change for phentermine to include a pediatric indication (down to age 10 years) and remove restrictions on the duration of use, thereby setting the stage for utilization in the primary care setting.

ELIGIBILITY:
Inclusion Criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female, aged 10-<18 years
* BMI ≥ 95th age- and sex-specific Centers for Disease Control (CDC) percentile
* Tanner stage ≥ 1
* Ability to take oral medication and be willing to adhere to the lifestyle therapy regimen

Exclusion Criteria:

* Contraindications to phentermine including: history of cardiovascular disease (including coronary artery disease, stroke, clinically significant congenital heart disease, clinically significant cardiac arrhythmias, congestive heart failure); glaucoma; current or recent (<14 days) use of MAO inhibitors; history of or current chemical dependency; current pregnancy or plans to be pregnant during course of study or lactation; known hypersensitivity to sympathomimetic amines.
* Hypertension
* Cardiac pacemaker
* Type 1 or type 2 diabetes mellitus
* Current or recent (<6 months prior to enrollment) use of weight loss medication(s)
* Current use of other sympathomimetic amines such as ADHD stimulants
* History of bariatric surgery
* Schizophrenia, psychosis, or mania
* Any history of suicide attempt
* Self-harm within 12 months prior to screening
* PHQ-9 score of ≥15 at screening
* Suicidal ideation of type 4 or 5 on C-SSRS in past month
* Hyperthyroidism

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change in body mass index (BMI) | 52 weeks
  To determine the effect of phentermine vs. placebo on body mass index reduction
Change in systolic and diastolic blood pressure | 52 weeks
  To determine the effect of phentermine vs. placebo on systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Change in triglyceride/HDL ratio | 52 weeks
  To determine the effect of phentermine vs. placebo on triglyceride and HDL levels in mg/dL
Change in inflammation | 52 weeks
  To determine the effect of phentermine vs. placebo on C-reactive protein in mg/L
Change in oxidative stress | 52 weeks
  To determine the effect of phentermine vs. placebo on oxidative LDL cholesterol in mg/dL
Change in Quality of Life | 52 weeks
  To determine the effect of phentermine vs. placebo on quality of life utilizing the Impact of Weight on Quality of Life-Kids (IWQOL). This questionnaire has four domains: physical comfort (6 items), body esteem (9 items), social life (6 items) and family relations (6 items). Scores range from 0 to 100, with 100 representing the best quality of life.

IPD SHARING:
Plan to Share IPD: Undecided